CLINICAL TRIAL: NCT00743652
Title: A Phase 3, Open Label Trial Evaluating the Safety, Immunogenicity and Impact of 13-valent Pneumococcal Conjugate Vaccine in Alaskan Native Children.
Brief Title: Study Evaluating the Impact of the 13-valent Pneumococcal Conjugate Vaccine (13vPnC) in Alaskan Native Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3010; B1851009
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2012-02-10 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Pneumococcal Disease; 13-valent Pneumococcal Vaccine
Keywords: 13 valent Pneumococcal Conjugate Vaccine; Antibody Response; safety; Alaskan Native Children
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group1 (Experimental): Subjects 6 weeks to <10 months of age with 0 prior dose of Prevnar.
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- Group 2 (Experimental): Subjects <12 months of age with 1 prior dose of Prevnar.
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- Group 3 (Experimental): Subjects <12 months of age with 2 prior doses of Prevnar.
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- Group 4 (Experimental): Subjects ≥12 months to <2 years of age.
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- Group 5 (Experimental): Subjects ≥2 years to <5 years of age
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 4 doses of 13vPnC (0.5ml, IM) will be administered. (3 doses infant series, and 1 toddler dose)
  Arms: Group1
Biological: 13-valent Pneumococcal Conjugate Vaccine — 3 doses of 13vPnC (0.5ml, IM) will be administered. (2 doses for infant series catch-up, and 1 toddler dose)
  Arms: Group 2
Biological: 13-valent Pneumococcal Conjugate Vaccine — 2 doses of 13vPnC (0.5ml, IM) will be administered. (1 dose infant series catch-up, and 1 toddler dose)
  Arms: Group 3
Biological: 13-valent Pneumococcal Conjugate Vaccine — 2 doses of 13vPnC (0.5ml, IM) will be administered. (2 catch-up dose(s) greater than 60 days apart )
  Arms: Group 4
Biological: 13-valent Pneumococcal Conjugate Vaccine — 1 dose of 13vPnC (0.5ml, IM) will be administered. (1 catch-up dose)
  Arms: Group 5

SUMMARY:
This study is to evaluate the safety, immunogenicity and impact of 13-valent Pneumococcal conjugate vaccine in Alaskan Native Children.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants 6 weeks to < 5years of age in good health, available for the entire study period and reachable by phone, parents able to complete all relevant study procedures.
* Infants who have received Prevnar are eligible to participate, but this is not required.
* Infants participating in the blood draws must live in a specific identified area (Yukon Kuskokwim Delta region)

Exclusion Criteria:

* Contraindication to vaccination with pneumococcal vaccine or allergic reaction to any vaccines or vaccine related components, immune deficiency, bleeding disorder or major known congenital malformation.

Ages: 42 Days to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (21):
  - Pfizer Investigational Site, Akiak, Alaska
  - Pfizer Investigational Site, Bethel, Alaska
  - Pfizer Investigational Site, Chefornak, Alaska
  - Pfizer Investigational Site, Chevak, Alaska
  - Pfizer Investigational Site, Eek, Alaska
  - Pfizer Investigational Site, Emmonak, Alaska
  - Pfizer Investigational Site, Hooper Bay, Alaska
  - Pfizer Investigational Site, Kalskag, Alaska
  - Pfizer Investigational Site, Kasigluk, Alaska
  - Pfizer Investigational Site, Kongiganak, Alaska
  - Pfizer Investigational Site, Kotlik, Alaska
  - Pfizer Investigational Site, Kwethluk, Alaska
  - Pfizer Investigational Site, Kwigillingok, Alaska
  - Pfizer Investigational Site, Mountain Village, Alaska
  - Pfizer Investigational Site, Napaskiak, Alaska
  - Pfizer Investigational Site, Newtok, Alaska
  - Pfizer Investigational Site, Nunapitchuk, Alaska
  - Pfizer Investigational Site, Russian Mission, Alaska
  - Pfizer Investigational Site, Scammon Bay, Alaska
  - Pfizer Investigational Site, Toksook Bay, Alaska
  - Pfizer Investigational Site, Tuluksak, Alaska

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3010&StudyName=Study%20Evaluating%20the%20Impact%20of%20the%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%20in%20Alaskan%20Native%20Children.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Blood sample was optional for subjects living in the Bethel area. Active vaccination stopped when 13-valent pneumococcal conjugate vaccine (13vPnC) was commercially available in Alaska. Study ended after a 6-month follow-up for safety following the last vaccination.
Groups:
- 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose): Participants 6 weeks to less than (<) 10 months of age with 0 prior doses of Prevnar received 3 single intramuscular (IM) 0.5 milliliter (mL) doses of 13-valent pneumococcal conjugate vaccine (13vPnC) at least 28 days apart (infant series), and a single IM 0.5 mL dose of 13vPnC at greater than (>) 12 months of age (toddler dose), at least 60 days after last infant dose.
- 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose): Participants <12 months of age with 1 prior dose of Prevnar received 2 single IM 0.5 mL doses of 13vPnC at least 28 days apart (infant series), and a single IM 0.5 mL dose of 13vPnC at >12 months of age (toddler dose), at least 60 days after last infant dose.
- 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose): Participants <12 months of age with 2 prior doses of Prevnar received a single IM 0.5 mL dose of 13vPnC (infant series) and a single IM 0.5 mL dose of 13vPnC at >12 months of age (toddler dose), at least 60 days after last infant dose.
- 13vPnC Group 4 (2 Catch-Up Doses): Participants greater than or equal to (≥) 12 months to <2 years of age received 2 single IM 0.5 mL doses of 13vPnC at least 60 days apart.
- 13vPnC Group 5 (1 Catch-Up Dose): Participants ≥2 years to <5 years of age received a single IM 0.5 mL dose of 13vPnC.
Period: Overall Study
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose) | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Started | 151 | 51 | 25 | 67 | 79
Vaccinated Dose 1 | 151 | 51 | 25 | 66 | 79
Vaccinated Dose 2 | 112 | 41 | 0 | 49 | 0
Vaccinated Dose 3 | 74 | 0 | 0 | 0 | 0
Toddler Dose | 15 | 23 | 16 | 0 | 0
Completed | 141 | 48 | 23 | 63 | 79
Not Completed | 10 | 3 | 2 | 4 | 0
Not completed — Parent/Legal Guardian Request | 3 | 2 | 2 | 2 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Investigator Request | 0 | 0 | 0 | 2 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose) | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose) | Total
Number analyzed (Participants) | 151 | 51 | 25 | 67 | 79 | 373
Age, Customized [Mean (Standard Deviation); unit: Months] | 1.4 (0.6) | 4.4 (0.8) | 7.1 (1.6) | 15.2 (3.4) | 40.1 (11.1) | 12.9 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 23 | 11 | 36 | 47 | 190
  Male | 78 | 28 | 14 | 31 | 32 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibody Level ≥0.35 Micrograms Per Milliliter (Mcg/mL) 1 Month After the Infant Series
Description: Percentage of participants in 13vPnC Groups 1, 2 and 3 achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: Evaluable immunogenicity population: received treatments as randomized at all expected doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations. N=number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 6 | 3
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotypes - serotype 6B | 100.0 [71.5 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 100.0 [71.5 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [29.2 to 100.0]
  Common serotypes - serotype 14 | 90.9 [58.7 to 99.8] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotype - serotype 19F | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotype - serotype 23F | 90.9 [58.7 to 99.8] | 83.3 [35.9 to 99.6] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 1 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 3 | 90.9 [58.7 to 99.8] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 5 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 6A | 90.9 [58.7 to 99.8] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 7F | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 19A | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]

2. Primary Outcome: Percentage of Participants Achieving Serotype-Specific Pneumococcal IgG Antibody Level ≥0.35 Mcg/mL 1 Month After the Toddler Dose
Description: Percentage of participants in 13vPnC Groups 1, 2, and 3 achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, and after vaccination 2 for Group 3.
Population: Evaluable immunogenicity population. N=number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 2
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 6B | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 14 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 19F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 23F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 1 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 3 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 5 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 6A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 7F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 19A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]

3. Primary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.35 Mcg/mL 1 Month After the Relevant Catch-Up Dose
Description: Percentage of participants in 13vPnC Groups 4 and 5 achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 9
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 6B | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 9V | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 14 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 18C | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 19F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 23F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 1 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 3 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 5 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 6A | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 7F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 19A | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]

4. Secondary Outcome: Percentage of Participants Achieving Serum IgG Antibody Level ≥0.35 Mcg/mL Prior to Vaccination With 13vPnC (Groups 4 and 5 Only)
Description: as for outcome 3
Time Frame: 28 to 56 days before vaccination 2 for Group 4, and before the single vaccination in Group 5.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 9
Percentage of Participants
  Common serotypes - serotype 4 | 50.0 [6.8 to 93.2] | 50.0 [15.7 to 84.3]
  Common serotypes - serotype 6B | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]
  Common serotypes - serotype 9V | 100.0 [39.8 to 100.0] | 66.7 [29.9 to 92.5]
  Common serotypes - serotype 14 | 100.0 [29.2 to 100.0] | 88.9 [51.8 to 99.7]
  Common serotype - serotype 18C | 75.0 [19.4 to 99.4] | 33.3 [7.5 to 70.1]
  Common serotype - serotype 19F | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]
  Common serotype - serotype 23F | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]
  Additional serotype - serotype 1 | 0.0 [0.0 to 60.2] | 12.5 [0.3 to 52.7]
  Additional serotype - serotype 3 | 0.0 [0.0 to 60.2] | 37.5 [8.5 to 75.5]
  Additional serotype - serotype 5 | 50.0 [6.8 to 93.2] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 6A | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]
  Additional serotype - serotype 7F | 0.0 [0.0 to 60.2] | 33.3 [7.5 to 70.1]
  Additional serotype - serotype 19A | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]

5. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥1.0 Mcg/mL 1 Month After the Infant Series
Description: Percentage of participants in 13vPnC Groups 1, 2, and 3 achieving predefined antibody threshold ≥1.0 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 6 | 3
Percentage of Participants
  Common serotypes - serotype 4 | 90.9 [58.7 to 99.8] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotypes - serotype 6B | 72.7 [39.0 to 94.0] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 81.8 [48.2 to 97.7] | 66.7 [22.3 to 95.7] | 66.7 [9.4 to 99.2]
  Common serotypes - serotype 14 | 90.9 [58.7 to 99.8] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 63.6 [30.8 to 89.1] | 83.3 [35.9 to 99.6] | 100.0 [29.2 to 100.0]
  Common serotype - serotype 19F | 100.0 [71.5 to 100.0] | 66.7 [22.3 to 95.7] | 100.0 [29.2 to 100.0]
  Common serotype - serotype 23F | 63.6 [30.8 to 89.1] | 50.0 [11.8 to 88.2] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 1 | 81.8 [48.2 to 97.7] | 83.3 [35.9 to 99.6] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 3 | 54.5 [23.4 to 83.3] | 66.7 [22.3 to 95.7] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 5 | 81.8 [48.2 to 97.7] | 83.3 [35.9 to 99.6] | 66.7 [9.4 to 99.2]
  Additional serotype - serotype 6A | 72.7 [39.0 to 94.0] | 83.3 [35.9 to 99.6] | 66.7 [9.4 to 99.2]
  Additional serotype - serotype 7F | 100.0 [71.5 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 19A | 72.7 [39.0 to 94.0] | 50.0 [11.8 to 88.2] | 33.3 [0.8 to 90.6]

6. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥1.0 Mcg/mL 1 Month After the Toddler Dose
Description: as for outcome 5
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, and after vaccination 2 for Group 3.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 2
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 50.0 [1.3 to 98.7]
  Common serotypes - serotype 6B | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 50.0 [1.3 to 98.7]
  Common serotypes - serotype 14 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 100.0 [15.8 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 19F | 100.0 [15.8 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 23F | 100.0 [15.8 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 1 | 100.0 [15.8 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 3 | 50.0 [1.3 to 98.7] | 66.7 [22.3 to 95.7] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 5 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 6A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 7F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 19A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]

7. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥1.0 Mcg/mL 1 Month After the Relevant Catch-up Dose
Description: Percentage of participants in 13vPnC Groups 4 and 5 achieving predefined antibody threshold ≥1.0 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 9
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 6B | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 9V | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 14 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 18C | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 19F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 23F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 1 | 100.0 [39.8 to 100.0] | 66.7 [29.9 to 92.5]
  Additional serotype - serotype 3 | 100.0 [39.8 to 100.0] | 77.8 [40.0 to 97.2]
  Additional serotype - serotype 5 | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]
  Additional serotype - serotype 6A | 100.0 [39.8 to 100.0] | 88.9 [51.8 to 99.7]
  Additional serotype - serotype 7F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 19A | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]

8. Secondary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Catch-up Dose 1
Description: Local reactions were reported by the parent/legal guardian using a diary card. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may have been represented in more than 1 category.
Time Frame: Day 1 through Day 7 after vaccination 1 for Group 4 and after the single vaccination in Group 5.
Population: Safety Population: all participants who received at least 1 dose of 13vPnC; N=number of participants reporting yes for at least 1 day or no for all days; n=number of participants with specific characteristic
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 65 | 77
Percentage of Participants
  Tenderness: Any (n=65,77) | 32.3 | 48.1
  Tenderness: Significant (n=63,77) | 3.2 | 9.1
  Swelling: Any (n=64,77) | 7.8 | 7.8
  Swelling: Mild (n=62,76) | 3.2 | 2.6
  Swelling: Moderate (n=63,77) | 3.2 | 6.5
  Swelling: Severe (n=63,77) | 1.6 | 2.6
  Redness: Any (n=65,77) | 15.4 | 13.0
  Redness: Mild (n=63,77) | 11.1 | 11.7
  Redness: Moderate (n=64,77) | 4.7 | 5.2
  Redness: Severe (n=63,77) | 1.6 | 2.6

9. Secondary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: Catch-up Dose 2
Description: as for outcome 8
Time Frame: Day 1 through Day 7 after vaccination 2 for Group 4
Population: Safety Population; N=number of participants reporting yes for at least 1 day or no for all days; n=number of participants with specific characteristic
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses)
Number analyzed (Participants) | 49
Percentage of Participants
  Tenderness: Any (n=49) | 36.7
  Tenderness: Significant (n=49) | 10.2
  Swelling: Any (n=48) | 10.4
  Swelling: Mild (n=47) | 8.5
  Swelling: Moderate (n=47) | 0.0
  Swelling: Severe (n=47) | 0.0
  Redness: Any (n=49) | 6.1
  Redness: Mild (n=48) | 4.2
  Redness: Moderate (n=48) | 0.0
  Redness: Severe (n=48) | 0.0

10. Secondary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Catch-up Dose 1
Description: Systemic events (any fever 38 degrees Celsius [C] or higher, decreased appetite, irritability, increased sleep, decreased sleep, hives [urticaria], and use of antipyretic medication) were reported using a diary card. Participants may have been represented in more than 1 category.
Time Frame: Day 1 through Day 7 after vaccination 1 for Group 4 and after the single vaccination in Group 5.
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 66 | 77
Percentage of Participants
  Fever ≥38 degrees C but ≤39 degrees C (n=35,47) | 42.9 | 27.7
  Fever >39 degrees C but ≤40 degrees C (n=29,43) | 20.7 | 11.6
  Fever >40 degrees C (n=28,40) | 7.1 | 0
  Decreased appetite (n=66,77) | 31.8 | 24.7
  Irritability (n=66,77) | 53.0 | 41.6
  Increased sleep (n=66,77) | 33.3 | 22.1
  Decreased sleep (n=66,77) | 24.2 | 11.7
  Hives (urticaria) (n=66,77) | 3.0 | 2.6
  Use of medication to treat symptoms (n=65,77) | 50.8 | 33.8

11. Secondary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: Catch-up Dose 2
Description: Systemic events (any fever 38 degrees C or higher, decreased appetite, irritability, increased sleep, decreased sleep, hives [urticaria], and use of antipyretic medication) were reported using a diary card. Participants may have been represented in more than 1 category.
Time Frame: Day 1 through Day 7 after vaccination 2 for Group 4
Population: as for outcome 9
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses)
Number analyzed (Participants) | 49
Percentage of Participants
  Fever ≥38 degrees C but ≤39 degrees C (n=26) | 23.1
  Fever >39 degrees C but ≤40 degrees C (n=22) | 9.1
  Fever >40 degrees C (n=21) | 0.0
  Decreased appetite (n=49) | 22.4
  Irritability (n=49) | 57.1
  Increased sleep (n=49) | 26.5
  Decreased sleep (n=49) | 4.1
  Hives (urticaria) (n=49) | 2.0
  Use of medication to treat symptoms (n=49) | 42.9

12. Other Pre Specified Outcome: Number of Cases of Invasive Pneumococcal Disease (IPD) in Participants Less Than 5 Years of Age Due to Any Serotype Contained in 13vPnC
Description: In order to assess the impact of 13vPnC on the incidence of IPD in the Yukon Kuskokwim (YK) Delta region, the Centers for Disease Control and Prevention (CDC) Arctic Investigation Program (AIP) accessed IPD data through evaluation of ongoing statewide IPD surveillance in Alaska. The CDC's AIP followed IPD (including serotype and vaccination history) to show whether identified cases of IPD received Prevnar, 13vPnC, or both. These data were combined with statewide data and used to identify the overall trend in IPD in the YK Delta region after introduction of 13vPnC.
Time Frame: Baseline to 6 months after last vaccination
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- 13vPnC (All Participants): All participants 6 weeks to <5 years of age who received at least one single IM 0.5 mL dose of 13vPnC in either the infant series or the toddler dose.
Arm/Group | 13vPnC (All Participants)
Number analyzed (Participants) | 373
Participants | 0

13. Other Pre Specified Outcome: Percentage of Participants Achieving Serotype-Specific Pneumococcal IgG Antibody Level ≥0.15 Mcg/mL 1 Month After the Infant Series
Description: Percentage of participants in 13vPnC Groups 1, 2, and 3 achieving predefined antibody threshold ≥0.15 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 6 | 3
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotypes - serotype 6B | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotypes - serotype 14 | 90.9 [58.7 to 99.8] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotype - serotype 19F | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Common serotype - serotype 23F | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 1 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 3 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 5 | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 6A | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 7F | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 19A | 100.0 [71.5 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [29.2 to 100.0]

14. Other Pre Specified Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.15 Mcg/mL 1 Month After the Toddler Dose
Description: as for outcome 13
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, and after vaccination 2 for Group 3.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 2
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 6B | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 14 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 19F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 23F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 1 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 3 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 5 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 6A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 7F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 19A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [15.8 to 100.0]

15. Other Pre Specified Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal IgG Antibody Level ≥0.15 Mcg/mL 1 Month After the Relevant Catch-up Dose
Description: Percentage of participants in 13vPnC Groups 4 and 5 achieving predefined antibody threshold ≥0.15 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based upon the observed proportion of participants.
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 9
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 6B | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 9V | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotypes - serotype 14 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 18C | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 19F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Common serotype - serotype 23F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 1 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 3 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 5 | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 6A | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 7F | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]
  Additional serotype - serotype 19A | 100.0 [39.8 to 100.0] | 100.0 [66.4 to 100.0]

16. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-Specific Pneumococcal IgG Antibodies 1 Month After the Infant Series
Description: Antibody GMCs (mcg/mL) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) with 2-sided 95% CIs were evaluated. CIs are back transformations of confidence levels based on Student t distribution for mean logarithm of concentrations. GMCs were calculated using all participants with available data for specified blood draw.
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: Evaluable immunogenicity population. N=number of participants with a determinate antibody concentration to the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 6 | 3
mcg/mL
  Common serotypes - serotype 4 | 2.64 [1.55 to 4.49] | 2.11 [0.93 to 4.80] | 4.27 [0.49 to 37.05]
  Common serotypes - serotype 6B | 2.74 [1.23 to 6.12] | 2.59 [0.55 to 12.26] | 28.60 [0.12 to 7043.76]
  Common serotypes - serotype 9V | 1.38 [0.97 to 1.98] | 1.04 [0.46 to 2.38] | 1.60 [0.31 to 8.37]
  Common serotypes - serotype 14 | 4.78 [1.71 to 13.33] | 4.08 [1.68 to 9.88] | 10.73 [0.06 to 1894.14]
  Common serotype - serotype 18C | 1.83 [1.04 to 3.21] | 1.66 [0.92 to 2.98] | 2.99 [0.40 to 22.62]
  Common serotype - serotype 19F | 3.55 [2.10 to 6.01] | 1.61 [0.65 to 4.01] | 2.37 [1.43 to 3.93]
  Common serotype - serotype 23F | 1.54 [0.79 to 3.01] | 1.03 [0.35 to 3.04] | 3.37 [1.18 to 9.66]
  Additional serotype - serotype 1 | 3.33 [1.68 to 6.62] | 3.02 [1.06 to 8.60] | 2.87 [0.30 to 27.24]
  Additional serotype - serotype 3 | 0.79 [0.51 to 1.22] | 1.61 [0.62 to 4.16] | 5.07 [1.53 to 16.79]
  Additional serotype - serotype 5 | 2.89 [1.57 to 5.31] | 1.93 [1.14 to 3.26] | 1.75 [0.25 to 12.25]
  Additional serotype - serotype 6A | 2.19 [0.93 to 5.16] | 2.48 [0.91 to 6.78] | 5.41 [0.01 to 2495.50]
  Additional serotype - serotype 7F | 3.34 [1.99 to 5.61] | 3.18 [1.24 to 8.12] | 6.21 [1.84 to 20.92]
  Additional serotype - serotype 19A | 1.87 [1.11 to 3.17] | 1.35 [0.56 to 3.25] | 0.97 [0.37 to 2.53]

17. Other Pre Specified Outcome: GMC for Serotype-Specific Pneumococcal IgG Antibodies 1 Month After the Toddler Dose
Description: Antibody GMCs (mcg/mL) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A). GMC (13vPnC) with 2-sided 95% CIs were evaluated. CIs are back transformations of confidence levels based on Student t distribution for mean logarithm of concentrations. GMCs were calculated using all participants with available data for specified blood draw.
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, after vaccination 2 for Group 3.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 2
mcg/mL
  Common serotypes - serotype 4 | 7.16 [0.00 to 199911.7] | 2.55 [1.44 to 4.53] | 1.76 [0.00 to 4004.84]
  Common serotypes - serotype 6B | 13.64 [0.00 to NA] — value=3.929*10^11 | 12.01 [4.23 to 34.08] | 11.32 [0.01 to 11544.32]
  Common serotypes - serotype 9V | 2.17 [0.01 to 373.79] | 2.20 [1.30 to 3.73] | 1.30 [0.00 to 2387.89]
  Common serotypes - serotype 14 | 12.18 [0.06 to 2411.14] | 11.42 [5.90 to 22.12] | 8.54 [0.19 to 377.53]
  Common serotype - serotype 18C | 2.35 [0.00 to 1681.49] | 2.22 [1.22 to 4.03] | 2.42 [0.08 to 72.55]
  Common serotype - serotype 19F | 11.00 [0.00 to 11762036] | 2.84 [1.03 to 7.79] | 3.65 [0.00 to 130178.5]
  Common serotype - serotype 23F | 3.79 [0.00 to 66245120] | 2.35 [0.88 to 6.27] | 3.96 [NA to NA] — n=2 for this serotype, and the value for both participants was 3.96, thus there was no variability so 95% CI could not be determined
  Additional serotype - serotype 1 | 2.15 [0.00 to 9338.28] | 4.19 [1.46 to 12.02] | 16.70 [0.00 to 5685164]
  Additional serotype - serotype 3 | 0.73 [0.00 to 276.18] | 1.32 [0.63 to 2.78] | 1.63 [1.19 to 2.23]
  Additional serotype - serotype 5 | 4.69 [0.00 to 36146.55] | 3.56 [1.96 to 6.46] | 5.85 [0.02 to 1606.11]
  Additional serotype - serotype 6A | 17.14 [0.00 to NA] — value=6.518*10^11 | 7.79 [3.00 to 20.21] | 3.24 [0.01 to 1555.15]
  Additional serotype - serotype 7F | 7.45 [0.47 to 117.40] | 5.55 [2.59 to 11.87] | 4.50 [0.05 to 440.58]
  Additional serotype - serotype 19A | 10.53 [2.63 to 42.07] | 3.21 [1.23 to 8.39] | 8.86 [0.00 to 8014211]

18. Other Pre Specified Outcome: GMC for Serotype-specific Pneumococcal IgG Antibodies 1 Month After the Relevant Catch-up Dose
Description: as for outcome 16
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 9
mcg/mL
  Common serotypes - serotype 4 | 4.16 [1.16 to 14.91] | 4.92 [1.94 to 12.50]
  Common serotypes - serotype 6B | 16.49 [4.31 to 63.06] | 22.94 [10.84 to 48.52]
  Common serotypes - serotype 9V | 3.22 [1.20 to 8.64] | 5.16 [2.34 to 11.37]
  Common serotypes - serotype 14 | 9.02 [2.18 to 37.29] | 16.99 [6.08 to 47.48]
  Common serotype - serotype 18C | 4.22 [2.22 to 8.05] | 5.08 [2.43 to 10.63]
  Common serotype - serotype 19F | 3.39 [0.78 to 14.78] | 6.45 [4.23 to 9.83]
  Common serotype - serotype 23F | 4.94 [1.82 to 13.41] | 5.41 [2.30 to 12.74]
  Additional serotype - serotype 1 | 9.37 [2.89 to 30.34] | 1.25 [0.64 to 2.46]
  Additional serotype - serotype 3 | 1.65 [1.13 to 2.40] | 1.91 [1.06 to 3.46]
  Additional serotype - serotype 5 | 4.51 [2.77 to 7.34] | 2.31 [1.41 to 3.78]
  Additional serotype - serotype 6A | 7.42 [1.77 to 31.06] | 4.46 [2.09 to 9.48]
  Additional serotype - serotype 7F | 8.81 [3.32 to 23.39] | 3.14 [1.93 to 5.08]
  Additional serotype - serotype 19A | 4.40 [2.96 to 6.54] | 5.61 [2.69 to 11.70]

19. Other Pre Specified Outcome: Percentage of Participants Achieving Opsonophagocytic Assay (OPA) Titers ≥Lower Limit of Quantitation (LLOQ) Measured 1 Month After the Infant Series
Description: Percentage of participants in 13vPnC Groups 1, 2, and 3 achieving OPA with 95% CI for serotypes 4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F, and 19A. Exact 2-sided CI based upon the observed proportion of participants. The LLOQ in titers for each serotype was: Pn001, 18; Pn003, 12; Pn004, 21; Pn005, 29; Pn06A, 37; Pn06B, 43, Pn7F, 210; Pn09V, 345; Pn014, 35; Pn18C, 31; Pn19A, 18; Pn19F, 48; and Pn23F, 13. Limit of detection (LOD) established as lowest titer possible in assay, which was 8. OPA titers below LLOQ set to 0.5*LOD for analysis.
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: Evaluable immunogenicity population. N=number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 5 | 3
Percentage of Participants
  Common serotypes - serotype 4 | 88.9 [51.8 to 99.7] | 75.0 [19.4 to 99.4] | 66.7 [9.4 to 99.2]
  Common serotypes - serotype 6B | 100.0 [66.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotypes - serotype 9V | 30.0 [6.7 to 65.2] | 0.0 [0.0 to 70.8] | 66.7 [9.4 to 99.2]
  Common serotypes - serotype 14 | 100.0 [54.1 to 100.0] | 75.0 [19.4 to 99.4] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 18C | 100.0 [59.0 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [15.8 to 100.0]
  Common serotype - serotype 19F | 88.9 [51.8 to 99.7] | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 97.5]
  Common serotype - serotype 23F | 88.9 [51.8 to 99.7] | 66.7 [9.4 to 99.2] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 1 | 60.0 [26.2 to 87.8] | 0.0 [0.0 to 60.2] | 33.3 [0.8 to 90.6]
  Additional serotype - serotype 3 | 90.9 [58.7 to 99.8] | 100.0 [47.8 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 5 | 70.0 [34.8 to 93.3] | 60.0 [14.7 to 94.7] | 33.3 [0.8 to 90.6]
  Additional serotype - serotype 6A | 90.0 [55.5 to 99.7] | 100.0 [47.8 to 100.0] | 100.0 [29.2 to 100.0]
  Additional serotype - serotype 7F | 100.0 [69.2 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [15.8 to 100.0]
  Additional serotype - serotype 19A | 80.0 [44.4 to 97.5] | 75.0 [19.4 to 99.4] | 100.0 [15.8 to 100.0]

20. Other Pre Specified Outcome: Percentage of Participants Achieving OPA Titers ≥LLOQ Measured 1 Month After the Toddler Dose
Description: Percentage of participants in 13vPnC Groups 1, 2 and 3 achieving OPA with 95% CI for serotypes 4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F, and 19A. Exact 2-sided CI based upon the observed proportion of participants. The LLOQ in titers for each serotype was: Pn001, 18; Pn003, 12; Pn004, 21; Pn005, 29; Pn06A, 37; Pn06B, 43, Pn7F, 210; Pn09V, 345; Pn014, 35; Pn18C, 31; Pn19A, 18; Pn19F, 48; and Pn23F, 13. Limit of detection (LOD) established as lowest titer possible in assay, which was 8. OPA titers below LLOQ set to 0.5*LOD for analysis.
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, and after vaccination 2 for Group 3.
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 1
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [15.8 to 100.0] | 50.0 [11.8 to 88.2] | 100.0 [2.5 to 100.0]
  Common serotypes - serotype 6B | 100.0 [15.8 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [2.5 to 100.0]
  Common serotypes - serotype 9V | 100.0 [15.8 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [2.5 to 100.0]
  Common serotypes - serotype 14 | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [2.5 to 100.0]
  Common serotype - serotype 18C | 100.0 [2.5 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [2.5 to 100.0]
  Common serotype - serotype 19F | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7] | 100.0 [2.5 to 100.0]
  Common serotype - serotype 23F | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [2.5 to 100.0]
  Additional serotype - serotype 1 | 100.0 [15.8 to 100.0] | 83.3 [35.9 to 99.6] | 100.0 [2.5 to 100.0]
  Additional serotype - serotype 3 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [2.5 to 100.0]
  Additional serotype - serotype 5 | 100.0 [15.8 to 100.0] | 66.7 [22.3 to 95.7] | 100.0 [2.5 to 100.0]
  Additional serotype - serotype 6A | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [2.5 to 100.0]
  Additional serotype - serotype 7F | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [2.5 to 100.0]
  Additional serotype - serotype 19A | 100.0 [15.8 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [2.5 to 100.0]

21. Other Pre Specified Outcome: Percentage of Participants Achieving OPA Titers ≥LLOQ Measured 1 Month After the Relevant Catch-up Dose
Description: Percentage of participants in 13vPnC Groups 4 and 5 achieving OPA with 95% CI for serotypes 4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F, and 19A. Exact 2-sided CI based upon the observed proportion of participants. The LLOQ in titers for each serotype was: Pn001, 18; Pn003, 12; Pn004, 21; Pn005, 29; Pn06A, 37; Pn06B, 43, Pn7F, 210; Pn09V, 345; Pn014, 35; Pn18C, 31; Pn19A, 18; Pn19F, 48; and Pn23F, 13. Limit of detection (LOD) established as lowest titer possible in assay, which was 8. OPA titers below LLOQ set to 0.5*LOD for analysis.
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 8
Percentage of Participants
  Common serotypes - serotype 4 | 100.0 [29.2 to 100.0] | 100.0 [63.1 to 100.0]
  Common serotypes - serotype 6B | 100.0 [29.2 to 100.0] | 100.0 [54.1 to 100.0]
  Common serotypes - serotype 9V | 100.0 [39.8 to 100.0] | 100.0 [54.1 to 100.0]
  Common serotypes - serotype 14 | 100.0 [15.8 to 100.0] | 100.0 [54.1 to 100.0]
  Common serotype - serotype 18C | 100.0 [29.2 to 100.0] | 100.0 [54.1 to 100.0]
  Common serotype - serotype 19F | 100.0 [29.2 to 100.0] | 100.0 [54.1 to 100.0]
  Common serotype - serotype 23F | 100.0 [29.2 to 100.0] | 100.0 [54.1 to 100.0]
  Additional serotype - serotype 1 | 100.0 [39.8 to 100.0] | 87.5 [47.3 to 99.7]
  Additional serotype - serotype 3 | 100.0 [39.8 to 100.0] | 100.0 [63.1 to 100.0]
  Additional serotype - serotype 5 | 100.0 [39.8 to 100.0] | 75.0 [34.9 to 96.8]
  Additional serotype - serotype 6A | 100.0 [39.8 to 100.0] | 87.5 [47.3 to 99.7]
  Additional serotype - serotype 7F | 100.0 [39.8 to 100.0] | 100.0 [63.1 to 100.0]
  Additional serotype - serotype 19A | 100.0 [39.8 to 100.0] | 100.0 [47.8 to 100.0]

22. Other Pre Specified Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) 1 Month After the Infant Series
Description: Antibody geometric mean titers as measured by OPA assay for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A). GMTs were calculated using all participants with available data for the specified blood draw. CIs for the GMTs are back transformations of confidence levels based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 5 | 3
Titers
  Common serotypes - serotype 4 | 123 [38.4 to 390.6] | 116 [3.1 to 4294.7] | 36 [0.3 to 4185.7]
  Common serotypes - serotype 9V | 20 [3.1 to 123.1] | 4 [NA to NA] — Within group, confidence intervals for serotypes for which participants all have the same titer value were not computed since variability cannot be estimated. | 120 [0.1 to 199619.2]
  Common serotype - serotype 19F | 151 [49.6 to 457.7] | 31 [0.7 to 1348.9] | 4 [NA to NA] — Within group, confidence intervals for serotypes for which participants all have the same titer value were not computed since variability cannot be estimated.
  Common serotype - serotype 23F | 299 [79.5 to 1124.8] | 81 [0.1 to 52488.1] | 566 [182.6 to 1755.9]
  Additional serotype - serotype 1 | 41 [9.2 to 183.5] | 4 [NA to NA] — Within group, confidence intervals for serotypes for which participants all have the same titer value were not computed since variability cannot be estimated. | 7 [0.5 to 109.4]
  Additional serotype - serotype 3 | 58 [28.9 to 117.7] | 82 [21.7 to 311.6] | 206 [66.1 to 639.0]
  Additional serotype - serotype 5 | 26 [9.6 to 72.3] | 18 [2.9 to 110.8] | 9 [0.3 to 234.2]
  Additional serotype - serotype 6A | 731 [182.2 to 2933.6] | 1069 [337.1 to 3390.4] | 984 [179.7 to 5383.5]
  Additional serotype - serotype 7F | 1396 [790.5 to 2467.0] | 1177 [692.5 to 2001.6] | 3485 [2308.5 to 5261.5]
  Common serotype - serotype 6B | 1280 [610.3 to 2683.5] | 1450 [370.4 to 5675.6] | 1790 [0.0 to 72147076]
  Common serotype - serotype 14 | 332 [98.0 to 1124.2] | 71 [3.3 to 1516.0] | 449 [0.1 to 2059598]
  Common serotype - serotype 18C | 868 [304.4 to 2475.0] | 452 [67.7 to 3023.6] | 906 [0.6 to 1340206]
  Additional serotype - serotype 19A | 58 [17.7 to 191.3] | 158 [2.5 to 9872.6] | 380 [0.0 to NA] — value=1.3309*10^8

23. Other Pre Specified Outcome: Pneumococcal OPA GMTs 1 Month After the Toddler Dose
Description: Antibody geometric mean titers as measured by OPA assay for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A). GMTs were calculated using all subjects with available data for the specified blood draw. CIs for the GMTs are back transformations of confidence levels based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, after vaccination 2 for Group 3.
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 1
Titers
  Common serotypes - serotype 4 | 599 [422.4 to 850.2] | 58 [2.6 to 1317.2] | 220 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Common serotypes - serotype 9V | 428 [68.2 to 2681.9] | 460 [35.0 to 6035.8] | 2765 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Common serotypes - serotype 14 | 775 [5.8 to 104290.7] | 551 [73.6 to 4120.2] | 779 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Common serotype - serotype 18C | 3311 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated. | 387 [14.8 to 10145.6] | 4316 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Additional serotype - serotype 1 | 46 [0.1 to 14754.5] | 66 [14.4 to 305.2] | 165 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Additional serotype - serotype 3 | 159 [0.2 to 141793.2] | 138 [60.9 to 313.7] | 402 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Additional serotype - serotype 5 | 87 [0.8 to 9175.7] | 30 [5.4 to 164.2] | 88 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Additional serotype - serotype 7F | 4590 [258.5 to 81484.1] | 1575 [810.3 to 3061.7] | 6105 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Additional serotype - serotype 19A | 1259 [210.3 to 7542.2] | 140 [22.7 to 860.3] | 427 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Common serotype - serotype 6B | 1565 [0.0 to NA] — value=2.4794*10^8 | 605 [17.1 to 21473.7] | 12470 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Common serotype - serotype 19F | 397 [0.0 to NA] — value=2.4862*10^8 | 73 [2.5 to 2087.3] | 532 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Common serotype - serotype 23F | 227 [0.0 to NA] — value=1.208*10^12 | 313 [30.6 to 3195.2] | 1660 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.
  Additional serotype - serotype 6A | 3207 [0.0 to NA] — value=1.9613*10^9 | 1688 [480.3 to 5929.3] | 6954 [NA to NA] — Within group, confidence intervals for serotypes with only 1 participant who had a determinate OPA antibody titer were not computed since variability cannot be estimated.

24. Other Pre Specified Outcome: Pneumococcal OPA GMTs 1 Month After the Relevant Catch-up Dose
Description: Antibody geometric mean titers as measured by OPA assay for 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). GMTs were calculated using all participants with available data for the specified blood draw. CIs for the GMTs are back transformations of confidence levels based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 8
Titers
  Common serotypes - serotype 4 | 594 [107.1 to 3295.5] | 1165 [261.1 to 5197.9]
  Common serotypes - serotype 6B | 7236 [3423.7 to 15294.0] | 6795 [795.9 to 58012.5]
  Common serotypes - serotype 9V | 2748 [457.9 to 16485.4] | 2979 [883.6 to 10040.5]
  Common serotypes - serotype 14 | 1159 [31.2 to 42979.5] | 1547 [347.4 to 6892.2]
  Common serotype - serotype 18C | 5910 [1824.6 to 19141.1] | 1871 [915.7 to 3824.2]
  Common serotype - serotype 19F | 1584 [463.4 to 5417.3] | 594 [84.8 to 4164.9]
  Common serotype - serotype 23F | 2870 [2572.2 to 3203.4] | 1240 [423.0 to 3632.5]
  Additional serotype - serotype 1 | 402 [285.8 to 564.7] | 62 [18.0 to 211.6]
  Additional serotype - serotype 3 | 218 [102.0 to 466.8] | 202 [136.0 to 299.3]
  Additional serotype - serotype 5 | 128 [15.9 to 1032.0] | 63 [13.3 to 302.2]
  Additional serotype - serotype 6A | 9067 [5187.0 to 15848.5] | 2292 [231.2 to 22724.0]
  Additional serotype - serotype 7F | 7776 [3701.3 to 16335.8] | 6086 [2680.9 to 13818.2]
  Additional serotype - serotype 19A | 815 [549.9 to 1206.8] | 400 [68.4 to 2344.7]

25. Other Pre Specified Outcome: Correlation of OPA and IgG Values for Each 13vPnC Serotype 1 Month After the Infant Series
Time Frame: 28 to 56 days after vaccination 3 for Group 1, after vaccination 2 for Group 2, and after vaccination 1 for Group 3.
Population: Correlative analysis output data are only available as figures and were not analyzed or presented statistically.
Measure: Number; unit: Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 11 | 5 | 3
Participants | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically. | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically. | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically.

26. Other Pre Specified Outcome: Correlation of OPA and IgG Values for Each 13vPnC Serotype 1 Month After the Toddler Dose
Time Frame: 28 to 56 days after vaccination 4 for Group 1, after vaccination 3 for Group 2, and after vaccination 2 for Group 3.
Population: Correlative analysis output data are only available as figures and were not analyzed or presented statistically.
Measure: Number; unit: Participants
Arm/Group | 13vPnC Group 1 (3 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 2 (2 Doses Infant Series and 1 Toddler Dose) | 13vPnC Group 3 (1 Dose Infant Series and 1 Toddler Dose)
Number analyzed (Participants) | 2 | 6 | 1
Participants | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically. | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically. | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically.

27. Other Pre Specified Outcome: Correlation of OPA and IgG Values for Each 13vPnC Serotype 1 Month After the Relevant Catch-up Dose
Time Frame: 28 to 56 days after vaccination 2 for Group 4, and after the single vaccination in Group 5.
Population: Correlative analysis output data are only available as figures and were not analyzed or presented statistically.
Measure: Number; unit: Participants
Arm/Group | 13vPnC Group 4 (2 Catch-Up Doses) | 13vPnC Group 5 (1 Catch-Up Dose)
Number analyzed (Participants) | 4 | 8
Participants | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically. | NA — Correlative analysis output data are only available as figures and were not analyzed or presented statistically.

ADVERSE EVENTS:
Time Frame: Randomization to 6 months after last vaccination
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Group 1 (Infant Series): Participants 6 weeks to <10 months of age with 0 prior doses of Prevnar received 3 single IM 0.5 mL doses of 13vPnC at least 28 days apart (infant series).
- Group 2 (Infant Series): Participants <12 months of age with 1 prior dose of Prevnar received 2 single IM 0.5 mL doses of 13vPnC at least 28 days apart (infant series)
- Group 3 (Infant Series): Participants <12 months of age with 2 prior doses of Prevnar received a single IM 0.5 mL dose of 13vPnC (infant series)
- Group 1 (Toddler Dose); Group 2 (Toddler Dose); Group 3 (Toddler Dose): Participants >12 months of age received a single IM 0.5 mL dose of 13vPnC at least 60 days after last infant dose (toddler dose)
- Group 4 (2 Catch-Up Doses): Participants ≥12 months to <2 years of age received 2 single IM 0.5 mL doses of 13vPnC at least 60 days apart.
- Group 5 (1 Catch-Up Dose): Participants ≥2 years to <5 years of age received a single IM 0.5 mL dose of 13vPnC.
Arm/Group | Group 1 (Infant Series) | Group 2 (Infant Series) | Group 3 (Infant Series) | Group 1 (Toddler Dose) | Group 2 (Toddler Dose) | Group 3 (Toddler Dose) | Group 4 (2 Catch-Up Doses) | Group 5 (1 Catch-Up Dose)
Serious Adverse Events (participants affected / at risk) | 21/151 | 2/51 | 1/25 | 0/15 | 0/23 | 2/16 | 3/66 | 0/79
Other Adverse Events (participants affected / at risk) | 11/151 | 4/51 | 1/25 | 0/15 | 0/23 | 0/16 | 1/66 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Infant Series) (N=151) | Group 2 (Infant Series) (N=51) | Group 3 (Infant Series) (N=25) | Group 1 (Toddler Dose) (N=15) | Group 2 (Toddler Dose) (N=23) | Group 3 (Toddler Dose) (N=16) | Group 4 (2 Catch-Up Doses) (N=66) | Group 5 (1 Catch-Up Dose) (N=79)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis haemophilus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic arthritis haemophilus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Infant Series) (N=151) | Group 2 (Infant Series) (N=51) | Group 3 (Infant Series) (N=25) | Group 1 (Toddler Dose) (N=15) | Group 2 (Toddler Dose) (N=23) | Group 3 (Toddler Dose) (N=16) | Group 4 (2 Catch-Up Doses) (N=66) | Group 5 (1 Catch-Up Dose) (N=79)
Pyrexia (General disorders) | 9 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crying (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.